CLINICAL TRIAL: NCT04833517
Title: REALITY Study: Analysis of a Prospective REgistry to Assess Outcome and Toxicity of Targeted RadionucLide TherapY in Patients With mCRPC in Clinical Routine.
Brief Title: Prospective REgistry of Targeted RadionucLide TherapY in Patients With mCRPC (REALITY Study)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universität des Saarlandes (Other)
Responsible Party: Principal Investigator, Samer Ezziddin, MD, Director, Dept. of Nuclear Medicine, Universität des Saarlandes
Other Study IDs: RNT-Prostate
Record Dates: First submitted 2021-03-31; First posted 2021-04-06 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Prostate Cancer Metastatic; Castration Resistant Prostatic Cancer; Advanced Prostate Carcinoma
Keywords: mCRPC; Radioligand Therapy; PSMA; PSMA-targeted Therapy; Radionuclide Therapy; Ra-223; Bone-targeted Radionuclide Therapy; Radioembolization; SIRT
MeSH Terms: conditions — Prostatic Neoplasms, Castration-Resistant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Lu177 PSMA RLT: Lutetium-177 prostate-specific membrane antigen (Lu177 PSMA) radioligand therapy (RLT) according to standard local protocol
- Ac225 PSMA RLT: Actinium-225 prostate-specific membrane antigen (Ac225 PSMA) radioligand therapy (RLT) according to standard local protocol
- Tandem Lu177 / Ac225 PSMA RLT: Combined Lu177 / Ac225 PSMA radioligand therapy according to standard local protocol
- Ra223 chloride: Bone-targeted Radium-223 (Ra223) radionuclide therapy in standard application
- Sm153 EDTMP: Bone-targeted Samarium-153 (Sm153) EDTMP radionuclide therapy in standard application
- Y90 microspheres: Radioembolization with yttrium-90 (Y90) microspheres, standard methodology
- Tb161 PSMA RLT: Terbium-161 prostate-specific membrane antigen (Tb161 PSMA) radioligand therapy (RLT) according to standard local protocol

SUMMARY:
This prospective registry aims to assess outcome and toxicity of targeted radionuclide therapies in patients with advanced prostate cancer in clinical routine. While the major investigated treatment modality is prostate-specific membrane antigen (PSMA)-targeted radioligand therapy, also other radionuclide therapies such as Ra223 and liver-directed radioembolization are included. The investigators believe that prospectively assessed long-term outcome data on implementation of radionuclide therapy, especially in the palliative setting of advanced mCRPC, help to better define the real benefits and risks of the respective treatment modalities for patients regarding survival and quality-of-life.

DETAILED DESCRIPTION:
Targeted radionuclide therapy is comprised of different modalities that may be applied in advanced prostate cancer, either targeting bone metastases (mainly using Radium-223), any site of metastases with PSMA-expression (ß- / alpha-emitter labelled radioligands) or loco-regionally applying internal radiation (Yttrium-90 microspheres) to metastatic liver disease. While in Germany, each form of treatment is used in clinical routine, data is sparse regarding the real benefits and risks of respective modalities, also when used in a sequential order. As an example, patients receiving Ra223 treatment may later undergo PSMA targeted radioligand therapy, with little data available on dependent response relationships or cumulative risks. Prospective assessment of outcomes and toxicities in a radionuclide therapy registry is apparently superior over retrospective analyses of selected patient populations.

The goal of the REALITY study is to gain a better understanding of the real-life clinical application of radionuclide therapies, with a focus on PSMA-targeted radioligand therapy in a high-volume treatment centre, and the impact of each treatment for patient outcome.

Based on primary and secondary outcome measures the potential prediction of treatment benefit by baseline patient and tumor characteristics, and early changes of biomarkers will be of interest.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form (Registry Study Inclusion Form)

Inclusion Criteria for PSMA RLT:

* sufficient tumoral PSMA expression defined as tracer uptake markedly higher than (physiologic) uptake in healthy liver tissue.
* sufficient bone marrow reserve: leukocytes ≥ 2 G/L, platelets > 75 × 109/L
* sufficient overall patient condition: Eastern Oncology Cooperative Group (ECOG) performance status ≤ 3

Exclusion Criteria:

* Inability or unwillingness to provide informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced castration-resistant prostate cancer, who receive radionuclide treatment including PSMA-targeted radioligand therapy, Radium-223 or other bone-targeted radionuclide therapy and liver-directed radioembolization.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
PSA response | up to 10 years
  Best PSA response and PSA response after 3 months from start of radionuclide therapy
PSA-PFS | up to 10 years
  PSA-based progression-free survival (PFS) according to PCWG3 criteria. From date of start of radionuclide therapy until documented and confirmed PSA-progression
OS | up to 10 years
  Overall survival. From date of start of radionuclide therapy until the date of death from any cause assessed
Toxicity (adverse events) | up to 10 years
  All toxicity occurring after start of radionuclide treatment will be registered according to the Common Terminology Criteria for Adverse Events (CTCAE version 4.03).
Toxicity-related discontinuation of radionuclide treatment | up to 10 years
  Rate of toxicity-related discontinuation of radionuclide therapy

SECONDARY OUTCOMES:
Conventional imaging response | up to10 years
  Response to radionuclide therapy based on conventional imaging according to RECIST 1.1
Molecular imaging response | up to 10 years
  Response to radionuclide therapy based on molecular imaging
Quality-of-life in patients receiving radionuclide therapy | up to 10 years
  Quality-of-life assessed from start of radionuclide treatment by EORTC QLQ-C30 questionaires
Pain control achieved by radionuclide therapy | up to 10 years
  Based on VAS-BPI patient questionaires from start of radionuclide treatment
Absorbed doses achieved by radionuclide therapy | up to 10 years
  Absorbed doses in Gy/GBq based on intra- / posttherapeutic dosimetry when available

CONTACTS AND LOCATIONS:
Overall Officials: Samer Ezziddin, MSc, MD, PhD, Principal Investigator — Universität des Saarlandes
Locations (1):
- Dept. of Nuclear Medicine, Saarland University, Homburg, Saarland, Germany

REFERENCES:
- [Derived] Bastian MB, Speicher T, Blickle A, Burgard C, Bastian JLD, Bartholoma M, Schaefer-Schuler A, Maus S, Ezziddin S, Rosar F. Tolerability of PSMA radioligand therapy in metastatic prostate cancer patients with baseline mild to moderate leukopenia. EJNMMI Res. 2025 Jul 6;15(1):82. doi: 10.1186/s13550-025-01280-0. PMID 40619537
- [Derived] Rosar F, Schuler J, Burgard C, Blickle A, Bartholoma M, Maus S, Petto S, Khreish F, Schaefer A, Ezziddin S. Efficacy and safety of rechallenge [177Lu]Lu-PSMA-617 RLT after initial partial remission in patients with mCRPC: evaluation of a prospective registry (REALITY study). Eur J Nucl Med Mol Imaging. 2024 Nov;51(13):4151-4162. doi: 10.1007/s00259-024-06825-4. Epub 2024 Jul 15. PMID 39008067
- [Derived] Rosar F, Burgard C, Rohloff LV, Blickle A, Bartholoma M, Maus S, Petto S, Schaefer-Schuler A, Ezziddin S. 225 Ac-PSMA-617 Augmentation in High-Risk mCRPC Undergoing 177 Lu-PSMA-617 Radioligand Therapy : Pilot Experience From a Prospective Registry. Clin Nucl Med. 2024 Jul 1;49(7):621-629. doi: 10.1097/RLU.0000000000005253. Epub 2024 May 21. PMID 38769643
- [Derived] Burgard C, Hein C, Blickle A, Bartholoma M, Maus S, Petto S, Schaefer-Schuler A, Ezziddin S, Rosar F. Change in total lesion PSMA (TLP) during [177Lu]Lu-PSMA-617 radioligand therapy predicts overall survival in patients with mCRPC: monocentric evaluation of a prospective registry. Eur J Nucl Med Mol Imaging. 2024 Feb;51(3):885-895. doi: 10.1007/s00259-023-06476-x. Epub 2023 Oct 27. PMID 37889298